CLINICAL TRIAL: NCT03371277
Title: Attributional Style Assessment in Patients With Parkinson's Disease Treated With Deep Brain Stimulation
Brief Title: Attributional Style and Parkinson's Disease
Acronym: ParkAIHQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PO17112
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2018-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1 (Experimental): patients with Parkinson's disease treated with deep brain stimulation.
  Interventions: Other: Medical visit for specific questionnaires
- Arm2 (Experimental): patients with Parkinson's disease treated without deep brain stimulation.
  Interventions: Other: Medical visit for specific questionnaires

INTERVENTIONS:
Other: Medical visit for specific questionnaires — Ambiguous Intentions Hostility Questionnaire (AIHQ) developed by Combs (2007)

SUMMARY:
Parkinson's disease (PD) is a common neurodegenerative disorder affecting 1-2% of the population over 65 years-old. In addition to the motor impairment characterized by resting tremor, bradykinesia, rigidity and postural instability, patients suffer with non-motor symptoms such as dysautonomia syndrome, sleep disturbances, depressive disorders, delusional disorders and cognitive disorders. Research and management of these non-motor symptoms is essential because these can be disabling and have a negative impact on the quality of life of patients. Among cognitive functions, social cognition is defined as the aspect that is dedicated to process social information for adaptive functioning. More specifically, it refers to an intricate set of higher-order neuropsychological domains that allow for adaptive behaviors in response to others. Four dimensions are usually included in this construct: theory of mind (ToM), emotion processing, social perception and social knowledge, and attributional style. Recently, different categories of social cognition have been studied in patients suffering from PD, such as the ToM or the recognition of facial emotions. Other aspects of social cognition that seem relevant in this population are still poorly studied; the attributional style is a cognitive bias defined as "the way we explain the causes of the positive or negative events that occur". Indeed, different causes can be attributed to an event, and this attribution is shared between oneself, others and other factors related to the situation. People with attribution bias may mistakenly attribute to one cause all the situations. For example, when an individual blame the others for an event, he may develop a feeling of hostility that may lead to maladaptive behavior such as aggression and thus affect his social functioning. The impact of PD treatments, particularly deep brain stimulation (DBS), on the ToM has been studied, showing a deficit after stimulation. No study has assessed the impact of therapeutics on the attributional style of PD patients. In this context, it seems relevant to evaluate the effect of deep brain stimulation on the attributional style in this population.

DETAILED DESCRIPTION:
To explore attribution bias in PD population, the Ambiguous Intentions Hostility Questionnaire (AIHQ) developed by Combs (2007) will be used. The participants will be asked to read 15 vignettes, to imagine the scenario happening to her or him (e.g., ''You walk past a bunch of teenagers at a mall and you hear them start to laugh''), and to write down the reason why the other person (or persons) acted that way toward you. Two independent raters will subsequently code this written response for the purpose of computing a ''hostility index'' (described below). The participant will then rate, on Likert scales, whether the other person (or persons) performed the action on purpose (1 ''definitely no'' to 6 ''definitely yes''), how angry it would make them feel (1 ''not at all angry'' to 5 ''very angry''), and how much they would blame the other person (or persons) (1 ''not at all'' to 5 ''very much''). Finally, the participant will be asked to write down how she or he would respond to the situation, which will be later coded by two independent raters to compute an ''aggression index'' (described in Combs, 2007).

Socio-demographic data, subsyndromic symptoms of depression and anxiety, paranoia symptoms and cognitive functions will also be assessed to explore the confounding factors.

ELIGIBILITY:
Inclusion criteria :

* Diagnostic of Parkinson's disease by a neurologist
* Native French speaker
* Affiliated to social security
* Unmodified PD treatment for at least 2 weeks before the inclusion
* Over 18 years-old
* Accepting the study after reading the information note and signing the consentment form

Exclusion criteria :

* Diagnostic of bipolar disorder or schizophrenia
* Abuse and dependence on psychoactive substances according to the DSM V criteria
* Disabling sensory disorders
* Mental retardation or cognitive deterioration (e.g. dementia), with the incapacity to answer to the questionnaires.
* Patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-07-07 (Actual); Study Completion 2018-07-07 (Actual)

PRIMARY OUTCOMES:
Attributional style | Day 0
  The Ambiguous Intentions Hostility Questionnaire (Combs et al., 2006) will be used to assess attributional style

SECONDARY OUTCOMES:
depression | Day 0
  The Hamilton Depression Rating scale (Hamilton, 1967 )will be used to assess presence of depression

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Decombe L, Henry A, Decombe R, Tir M, Doe de Maindreville A, Galland Hairabedian L, Kaladjian A, Raucher-Chene D. "Accidental, really?" Attributional bias in patients with Parkinson's disease. Parkinsonism Relat Disord. 2022 Feb;95:18-22. doi: 10.1016/j.parkreldis.2021.12.013. Epub 2021 Dec 23. PMID 34959046